CLINICAL TRIAL: NCT02513680
Title: Effects of Application LED Therapy and Laser Therapy in Facial Rejuvenation: Pilot Study
Brief Title: Effects of Application LED Therapy and Laser Therapy in Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Patricia Viana da Rosa, Adjunct Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36980514.0.0000.5345
Record Dates: First submitted 2015-06-30; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Aging; Wrinkles
Keywords: Skin Aging; laser phototherapy; Rejuvenation; Infrared Rays/therapeutic use; Female; Humans; Esthetics; Phototherapy; facial rejuvenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LASER and LED therapy application (Active Comparator): The first group will use the two techniques under study combined: Infrared Laser + Amber LED (830 nm - 150mW + 590 nm - 1.500 mW)
  Interventions: Device: Infrared Laser + Amber LED
- LED Therapy application (Active Comparator): The second group will use only Amber LED (590 nm - 1.500 mW)
  Interventions: Device: Amber LED

INTERVENTIONS:
Device: Infrared Laser + Amber LED — This group will make the application on the machine program that uses laser and led together to photorejuvenation . Laser is applied for 30 seconds and soon after begins the LED by 2:30 minutes in each region to apply.
  Arms: LASER and LED therapy application
Device: Amber LED — This group will make the application on the machine program that uses LED photorejuvenation only 3 minutes of time for each area to be applied.
  Arms: LED Therapy application

SUMMARY:
In today's society, the search for keeping up with the appearance with no visible signs of aging has become common. Therefore, many therapies to try to mitigate these senility markers are present in specialized clinics. Such therapies seek grounding in the theories of how the skin and its appendages respond to the aging process, causing this way, they can be created ways to slow or minimize wrinkles and other consequences of this natural biological process. However, this process can be accelerated by exposure to ultraviolet light such as to toxic substances as well as tobacco, among others. The low-power laser and light emitted diode (LED) characterized by being non-ablative light source, which means phototherapy which does not cause physical damage to the epidermis, as the case of CO2 laser ablative and other methods. This study has the purpose of comparing the effects of combined application of low level laser with LED and LED action alone in facial rejuvenation. For this, the analysis of these effects will be conducted through digital photography, blinded assessment and customer satisfaction questionnaire.

DETAILED DESCRIPTION:
This is a pilot study seen the lack of studies on the subject chosen for a sample calculation accurately be defined. This will be done by 32 volunteers, respecting the criteria for inclusion and exclusion previously cited by reading and signing the Informed Consent and Clarified. The sample comprises a total of 30 subjects, divided randomly into two groups with 16 subjects in each. The first group will make use of both techniques in combined study: Infrared Laser and Led Amber. The second group, in turn, will use only the Led Amber.These will be allocated randomly and intervention will be simple blind.They will be held 10 sessions in individual applications, both group 1 (Laser and LED) and group 2 (LED) and applications for two groups will occur once per week. Group 1 will make the application of the two techniques on the same day session. Both will be applied in the following areas of the face: chin / perioral, nasolabial folds, periorbital, frontal and glabellar region. Both groups act as their own controls before starting the sessions, to ensure that the changes observed in the skin is caused by the treatment of fact and not the environment. For this, the volunteers will be accompanied during the first month, with completion of a photograph at the beginning of the month to another month-end, as well as a questionnaire at the end of 30 days.

To monitor the results, will be held 4 shoots of the subjects in the study. The first session will take place at the first meeting with the patients, who will undergo a 4-week follow-up without using any methodology. After these four weeks, a new shoot will be held to determine whether the environment was able to promote changes in the skin of patients or not. After this, it will start to bare-sessions. After five sessions of treatment, a new picture for monitoring will be held, and repeated this procedure at the end of treatment for so yes, compare the images and get search results.

To carry out the photos, there will be a standard procedure in order to maintain quality, the angle and the light always the same, so that the results observed can be truthful fact. Initially, the face of the patient will be cleaned, particularly aiming at the removal of cosmetic and excess oil on the surface to be photographed. This will precede the photographic record in at least 5 minutes so that friction marks and flushing fall apart.

Afterwards, the patients with the prisoners hair (or using burrows), will be photographed standing in front and lateral planes (both sides), parallel to the plane of the camera sensor. To better guide them, will be applied on the floor marks with the positions of the feet, to be followed.A camera mounted on the tripod, level and horizontal position, with the 105mm lens will be placed in proper height for framing the mouth, forehead and brows. The framework of each area will follow the alignment of facial landmarks to the camera's viewfinder grid in live view mode.

To photograph the brow area both iris will be aligned with the intersections between the line dividing the room and the lower horizontal lines that divide the extreme vertical side rooms of the grid. To shoot the mouth area "Cheilion" the two points will be aligned respectively with the intersections between the line that bisects the grid and the lines that divide the extreme horizontal side rooms. To photograph the area of the forehead (both sides) and the "Exocanthion" and "Otobasion Superious" points will be aligned with the intersections between the line that bisects the grid and the lines that divide the extreme horizontal side rooms. The flash is mounted on the hot shoe of the camera, set in TTL mode with the driven diffuser and will have its head directed forward. The camera will be displayed in manual mode, with f5.6 aperture, shutter speed to 1/60 second and 200 ISO.

At the end of the collection and collation, registration and randomization of the obtained photographs, there will be the evaluation of research students, who will receive the photos in random order and will have to put them in expected development order for a rejuvenation treatment. After learning the correct order, there will quantify the improvements in fine lines of the four areas chosen for analysis. In addition, two blind evaluators will be invited to participate in the project by analyzing the same way that researchers students. The external evaluators will be the ones who will have knowledge of what method the person was exposed. The evaluator will not know whether or not a placebo group in the study. Still, it is important to consider that the designated evaluator will be a person with extensive knowledge about the skin and possible treatments the same, so you can see exactly if there were no improvements or the skin of the participants. The analysis of the photos will take place in three steps:

STEP 1:

Slides with 3 or 4 photographs of each subject in random order (black and white photographs to color hair, earrings, not to interfere in the result).

The evaluator should classify the images in the order of 1-4, with 1 being the worst picture, and 4 the best (relative expression lines, skin texture and brightness) (it is expected that the treatment has left the skin better, so this sort order).

They will be received 4 slides pertaining to each subject, each containing the pictures of the respective regions assessed: frontal, nasolabial, periorbital, glabellar. Along with this, evaluators will be delivered to a table so that they can put the sort order of 1-4 each presented slide.

STEP 2:

Slide with a picture before starting treatment and the final photograph arranged chronologically (photographs in black and white).

The assessor should note the first and last picture of each region of each treated patient (4 regions per patient) and classify the changes in one of the degrees of the scale below:

0% = no change regarding the improvement of fine lines / wrinkles.

1% - 25% = little change regarding the improvement of fine lines / wrinkles, difficult to observe 25-50% = there has been a change regarding the improvement of fine lines / wrinkles, but nothing extremely significant 50% or more = a change in relation to improvement of fine lines / wrinkles is visible, the skin really improved considerably

STEP 3:

Slides containing two images of each patient in a more central area of the face (Vintage Photography).

The evaluator will receive the slides containing a photograph before the start of treatment and the last shot of each volunteer performed relating to a face of the central region. It is the evaluator understand the following items:

1. Voluntary skin had spots? Yes or no?
2. If stains showed there was a difference in the amount (uniformity) of the skin before and after treatment? Yes or no?

In addition, throughout this study of customer satisfaction questionnaires will be carried out in order to monitor whether the patient is enjoying the treatment, it is believed that is actually running (sorting qualitivamente the improvement of fine lines) and recommend this to other people.Thus, the treatment becomes, in general, valuable, since it is known that on the market, the transmission from one person to another feature of procedures that results is an efficient form of this disclosure. Such tests will be done in the middle of treatment (5 sessions) and at the end of it (10 sessions) to compare whether there was a change of the view in the meantime.

ELIGIBILITY:
Inclusion Criteria:

* Female patients study present ages 30 and 50;
* Wrinkles compatible with the G2 and G3 stages measured according Glogau scale;
* Phototypes consistent with those described and between FZ1 to FZ4 according to Fitzpatrick scale;
* Patients without previous hypersensitivity reaction
* Patients must agree and sign the consent form and clarified.

Exclusion Criteria:

* Patients who present wrinkles compatible with the G1 and G4 stages of Glogau scale;
* Patients who present FZ5 and FZ6 phototypes according to Fitzpatrick scale to increase the risk of burns from the treatment.
* Patients who have experienced any hypersensitivity reaction in some prior treatment has been paid;
* Volunteers who are being subjected to treatments with acids synthesized from vitamin A ( acid retinoic , Retinol A, Vitanol A, Retin , Isotretinoin , tretinoin ) and Vitamin C (creams , serums , capsules ) and / or tetracycline and / or which have made facial aesthetic treatments

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy of LED and Laser therapy in facial photorejuvenation | Ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lívia S Born, Principal Investigator — Federal University of Health Science of Porto Alegre; Ana Claudia Fedi, Principal Investigator — Federal University of Health Science of Porto Alegre